CLINICAL TRIAL: NCT02739763
Title: Controlled Human Malaria Infection (CHMI) to Assess Human Immunity to P. Falciparum Using Sporozoites Administered by Direct Venous Inoculation
Brief Title: Controlled Human Malaria Infection in Semi-Immune Kenyan Adults. (CHMI-SIKA)
Acronym: CHMI-SIKA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: KEMRI-Wellcome Trust Collaborative Research Program (Other); Sanaria Inc. (Industry); KEMRI Centre for Clinical Research (Unknown); Pwani University (Unknown); University of Cambridge (Other); Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OXTREC 2-16; KEMRI/CGMRC/CSC/029/2015 (Other: KEMRI Scientific and Ethics Review Unit)
Record Dates: First submitted 2016-04-13; First posted 2016-04-15 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Malaria
Keywords: PfSPZ; Semi-immune adults; Kenya; challenge; CHMI; malaria
MeSH Terms: conditions — Malaria | interventions — thrombospondin-related adhesive protein, protozoan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plasmodium falciparum sprozoite (PfSPZ) challenge (Experimental): Challenge agent
  Interventions: Biological: Plasmodium falciparum sporozoite (PfSPZ)

INTERVENTIONS:
Biological: Plasmodium falciparum sporozoite (PfSPZ) — Plasmodium falciparum sporozoites

SUMMARY:
The investigators wish to understand how resistance to malaria develops and how this affects the growth rate of malaria in individuals who have past exposure to malaria.

DETAILED DESCRIPTION:
Malaria remains a major public health threat despite regulatory approval of a partially effective pre-erythrocytic malaria vaccine. There is an urgent need to accelerate the development of a more effective multi-stage vaccine. Controlled human malaria infection (CHMI) has been shown to be an important tool for the assessment of the efficacy of novel malaria vaccines and drugs prior to field trials. CHMI also allows for the evaluation of immunity to malaria and parasite growth rates in vivo. This is particularly useful in individuals from endemic areas with a level of exposure and immunity to malaria. Thus CHMI in individuals with prior exposure to malaria could be a valuable tool to accelerate malaria vaccine development. In this study, the investigators aim to use CHMI in semi-immune adults to provide a comprehensive prioritization of antigens associated with blood-stage immunity for vaccine development. The investigators will comprehensively characterize immunity to malaria using >100 antigens in up to 2,000 semi-immune adults, from known areas of malaria endemicity in Kenya, then select 200 individuals with a range of different immunological profiles, and conduct CHMI studies with serial quantitative polymerase chain reaction (PCR) to measure the parasite growth rate in vivo and relate this to host immunity. This will also involve analysing the relationship with functional immunity assessed by laboratory assays.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Informed consent.
* Use of effective method of contraception for duration of study (women only). The investigators will ask the female volunteers to come with their family planning records to verify. Effective contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly, in accordance with the product label. Examples of these include: combined oral contraceptives; injectable progestogen; implants of etenogestrel or levonorgestrel; intrauterine device or intrauterine system; male partner sterilisation at least 6 months prior to the female subject's entry into the study, and the relationship is monogamous; male condom combined with a vaginal spermicide (foam, gel, film, cream or suppository); and male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository).

Exclusion Criteria:

* Use of systemic antibiotics with known antimalarial activity within 30 days of administration of PfSPZ Challenge (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin).
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Current participation in another clinical trial or recent participation within 12 weeks of enrolment.
* Prior receipt of an investigational malaria vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* Any serious medical condition reported or identified during screening that increases the risk of CHMI.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination.
* Women only; pregnancy, or an intention to become pregnant during the duration of the study.
* Confirmed parasite positive by PCR a day before challenge i.e. at C-1.

Exclusion Criterion on Day of Challenge:

• Acute disease, defined as moderate or severe illness with or without fever (temperature >37.5°C).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-01 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Infectivity of PfSPZ (malaria infection) as determined by quantitative PCR | day 7 to day 21

SECONDARY OUTCOMES:
Safety profile of PfSPZ challenge via direct venous injection | day 0 to day 21
Parasite growth rates with respect to antibody responses to over 100 falciparum antigens | day 7 to day 21

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bejon, MD,PhD, Principal Investigator — KEMRI Wellcome Trust Research Programme and University of Oxford
Locations (2):
- Kenya (2):
  - KEMRI Wellcome Trust Research Programme, Kilifi, Coast
  - KEMRI Centre for Clinical Research, Nairobi, Nairobi County

IPD SHARING:
Plan to Share IPD: Yes
Study information will be made available through an open repository. The information to be made available will be anonymized so that there is no link to participants and will include data on antibody responses, parasite growth rates and any other data generated from samples obtained in this study, both generated from this current protocol or any future studies which will require additional ethical approval.

REFERENCES:
- [Derived] Kariuki SN, Macharia AW, Makale J, Nyamu W, Hoffman SL, Kapulu MC, Bejon P, Rayner JC, Williams TN; CHMI-SIKA Study Team. The Dantu blood group prevents parasite growth in vivo: Evidence from a controlled human malaria infection study. Elife. 2023 Jun 13;12:e83874. doi: 10.7554/eLife.83874. PMID 37310872
- [Derived] Li K, Tsukasa Y, Kurio M, Maeta K, Tsumadori A, Baba S, Nishimura R, Murakami A, Onodera K, Morimoto T, Uemura T, Usui T. Belly roll, a GPI-anchored Ly6 protein, regulates Drosophila melanogaster escape behaviors by modulating the excitability of nociceptive peptidergic interneurons. Elife. 2023 Jun 13;12:e83856. doi: 10.7554/eLife.83856. PMID 37309249
- [Derived] Musasia FK, Nkumama IN, Frank R, Kipkemboi V, Schneider M, Mwai K, Odera DO, Rosenkranz M, Furle K, Kimani D, Tuju J, Njuguna P, Hamaluba M, Kapulu MC, Wardemann H; CHMI-SIKA Study Team; Osier FHA. Phagocytosis of Plasmodium falciparum ring-stage parasites predicts protection against malaria. Nat Commun. 2022 Jul 14;13(1):4098. doi: 10.1038/s41467-022-31640-6. PMID 35835738
- [Derived] Kapulu MC, Kimani D, Njuguna P, Hamaluba M, Otieno E, Kimathi R, Tuju J, Sim BKL; CHMI-SIKA Study Team. Controlled human malaria infection (CHMI) outcomes in Kenyan adults is associated with prior history of malaria exposure and anti-schizont antibody response. BMC Infect Dis. 2022 Jan 24;22(1):86. doi: 10.1186/s12879-022-07044-8. PMID 35073864
- [Derived] Kapulu MC, Njuguna P, Hamaluba M, Kimani D, Ngoi JM, Musembi J, Ngoto O, Otieno E, Billingsley PF; Controlled Human Malaria Infection in Semi-Immune Kenyan Adults (CHMI-SIKA) Study Team. Safety and PCR monitoring in 161 semi-immune Kenyan adults following controlled human malaria infection. JCI Insight. 2021 Sep 8;6(17):e146443. doi: 10.1172/jci.insight.146443. PMID 34264864
- [Derived] Kapulu MC, Njuguna P, Hamaluba MM; CHMI-SIKA Study Team. Controlled Human Malaria Infection in Semi-Immune Kenyan Adults (CHMI-SIKA): a study protocol to investigate in vivo Plasmodium falciparum malaria parasite growth in the context of pre-existing immunity. Wellcome Open Res. 2019 Nov 14;3:155. doi: 10.12688/wellcomeopenres.14909.2. eCollection 2018. PMID 31803847